CLINICAL TRIAL: NCT00608621
Title: Influence of Physostigmine on Patient-Controlled Analgesia (PCA) in Postoperative Intensive Care Patients, Considering Pain Score, Opioid Consumption, Hemodynamics and Cognitive Function
Brief Title: Influence of Physostigmine on Patient-Controlled Analgesia (PCA) in Postoperative Intensive Care Patients
Acronym: ANA06103
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Collaborators: University of Mannheim (Other)
Responsible Party: Klinikum Ludwigshafen, Dep. of Anesthesiology, Dr. K. D. Röhm
Other Study IDs: ANA06103
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2007-12

CONDITIONS: Pain
Keywords: physostigmine; postoperative analgesia; pain; patient-controlled analgesia; Opioid consumption; Pain quality (VAS Score); Hemodynamics; Mobilisation; Side effects
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-physostigmine: Physostigmine 4 mg in 50 ml NaCl 0.9% per 24 h as syringe pump continuously for 48 hours, plus physostigmine 2mg (in NaCl 0.9% 50 ml)at termination of sedation
  PCA: Patient-controlled analgesia with piritramide 1 mg/ml, on demand: bolus of 2 mg, maximum of 10 mg in 60 min
- 2-placebo: NaCl 0.9% 50 ml per 24 h continuously over 48 hours, plus 50 ml NaCl 0.9% at termination of sedation
  PCA: Patient-controlled analgesia with piritramid 1 mg/ml, on demand: bolus of 2 mg, maximum of 10 mg in 60 min

SUMMARY:
The study is to evaluate the influence of physostigmine in the postoperative period in intensive care patients considering pain quality, opioid consumption, hemodynamics and mobilisation.

DETAILED DESCRIPTION:
Pain management is of major concern in the postoperative period, mostly based on opioids. In numerous experimental and clinical trials cholinergic mechanisms have been demonstrated to play an important antinociceptive role. Physostigmine, a central cholineresterase inhibitor, has been shown to produce analgesia and enhance opiate analgesia after systemic injection. This action is not based on µ-receptor (opioid) activity, but can be mostly explained by stimulation of serotonine (5-HT-3) receptors. The major withdrawal of utilizating physostigmine in postoperative care, is due to its short duration of action.

In the present study, we examined the effect of a continuous intavenous physostigmine application during a patient-controlled analgesia with piritramide for 48 hours compared to a placebo infusion with NaCl.

Major concern was set for consumption of analgesics, VAS-pain scale, hemodynamics, mobilisation and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Indication for postoperative pain therapy and admission to ICU
* ASA I-III
* Weight 50-125 kg
* Patients that are willing to participate in the present study

Exclusion Criteria:

* Peridural anesthesia for pain management
* Severe left ventricular function (EF <30%)
* Severe/exacerbated COPD; Asthma
* ASA IV-V
* Chronic renal insufficiency(Creatinine > 1,5 mg/dl)
* Ulcera ventriculi
* Known allergy to any of the study agents
* Hb preoperative <9,5 g/dl
* Alcohol,drug and/or tablet abuse (Opioids, NSAR)
* Emergency operation
* Pregnancy
* Women of childbearing age and without a negative pregnancy test
* Severe liver disease (GOT oder GPT > 45 U/L)
* Severe neurologica derangements (e.g. M. Parkinson, Multiple Sklerosis)
* History of apoplexia <6 Monate or residua
* Perioperative myocardial infarction
* Patients that are not able to agree to the present study
* Patients that refuse to participate in the present study
* Patients that are part of any other study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective major surgery, postoperative ICU patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 48 hours

SECONDARY OUTCOMES:
pain quality (VAS) mobilisation hemodynamics side effects | operation to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Konrad, Prof., Principal Investigator — University Hospital Mannheim, Department of Anesthesiology; Kerstin D. Roehm, MD, Study Director — Klinikum Ludwigshafen, Department of Anesthesiology
Locations (1):
- Klinkum Ludwigshafen, Department of Anesthesiology, Ludwigshafen, Germany

REFERENCES:
- [Background] Beilin B, Bessler H, Papismedov L, Weinstock M, Shavit Y. Continuous physostigmine combined with morphine-based patient-controlled analgesia in the postoperative period. Acta Anaesthesiol Scand. 2005 Jan;49(1):78-84. doi: 10.1111/j.1399-6576.2004.00548.x. PMID 15675987
- [Background] Rohm KD, Riechmann J, Boldt J, Schollhorn T, Piper SN. Retracted: Do patients profit from physostigmine in recovery from desflurane anaesthesia? Acta Anaesthesiol Scand. 2007 Mar;51(3):278-83. doi: 10.1111/j.1399-6576.2006.01238.x. Epub 2007 Jan 23. PMID 17250745
- [Background] Aiello-Malmberg P, Bartolini A, Bartolini R, Galli A. Effects of morphine, physostigmine and raphe nuclei stimulation on 5-hydroxytryptamine release from the cerebral cortex of the cat. Br J Pharmacol. 1979 Apr;65(4):547-55. doi: 10.1111/j.1476-5381.1979.tb07863.x. PMID 435680
- [Background] Passchier J, Rupreht J, Koenders ME, Olree M, Luitwieler RL, Bonke B. Patient-controlled analgesia (PCA) leads to more postoperative pain relief, but also to more fatigue and less vigour. Acta Anaesthesiol Scand. 1993 Oct;37(7):659-63. doi: 10.1111/j.1399-6576.1993.tb03784.x. PMID 8249554
- [Background] Rupreht J, Schneck HJ, Dworacek B. [Physostigmine--recent pharmacologic data and their significance for practical use]. Anaesthesiol Reanim. 1989;14(4):235-41. German. PMID 2675888